CLINICAL TRIAL: NCT05251727
Title: Double-blind, Placebo-controlled, Randomized, Dose-escalating, Multi-center, Phase 1 Study to Assess the Safety and Tolerability of ART-123 With Leucovorin/5-fluorouracil/Oxaliplatin and Bevacizumab in Metastatic Colorectal Cancer Patients
Brief Title: Assess Safety and Tolerability of ART-123 + FOLFOX + Bevacizumab in Metastatic Colorectal Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ART-123.PN101
Record Dates: First submitted 2022-01-07; First posted 2022-02-23 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — ART123

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Lowest Dose (Experimental): Lyophilized ART-123 reconstituted with sterile water for injection and administered by intravenous infusion over approximately 30 minutes prior to chemotherapy on Day 1 of cycle (for up to 3 cycles including bevacizumab)
  Interventions: Drug: thrombomodulin alfa
- Low Dose (Experimental): Lyophilized ART-123 reconstituted with sterile water for injection and administered by intravenous infusion over approximately 30 minutes prior to chemotherapy on Day 1 of cycle (for up to 3 cycles including bevacizumab)"
  Interventions: Drug: thrombomodulin alfa
- Medium Dose (Experimental): Lyophilized ART-123 reconstituted with sterile water for injection and administered by intravenous infusion over approximately 30 minutes prior to chemotherapy on Day 1 of cycle (for up to 3 cycles including bevacizumab)"
  Interventions: Drug: thrombomodulin alfa
- High Dose (Experimental): Lyophilized ART-123 reconstituted with sterile water for injection and administered by intravenous infusion over approximately 30 minutes prior to chemotherapy on Day 1 of cycle (for up to 3 cycles including bevacizumab)"
  Interventions: Drug: thrombomodulin alfa
- Highest Dose (Experimental): Lyophilized ART-123 reconstituted with sterile water for injection and administered by intravenous infusion over approximately 30 minutes prior to chemotherapy on Day 1 of cycle (for up to 3 cycles including bevacizumab)"
  Interventions: Drug: thrombomodulin alfa
- Placebo (Placebo Comparator): Lyophilized placebo reconstituted with sterile water for injection and administered by intravenous infusion over approximately 30 minutes prior to chemotherapy on Day 1 of cycle (for up to 3 cycles including bevacizumab)"
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: thrombomodulin alfa — Weight based dose of reconstituted treatment
  Other Names: ART-123
  Arms: High Dose; Highest Dose; Low Dose; Lowest Dose; Medium Dose
Drug: Placebo — Weight based dose of reconstituted treatment
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of ART-123 in patients with metastatic colorectal cancer who receive oxaliplatin-containing chemotherapy and bevacizumab

DETAILED DESCRIPTION:
To compare the safety and tolerability of ART-123 to placebo in patients with metastatic colorectal cancer who receive oxaliplatin-containing chemotherapy and bevacizumab

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Metastatic colorectal cancer; pathologically confirmed adenocarcinoma of the colon or rectum
* ECOG performance status of 0 or 1
* The most recent laboratory findings (including for liver and kidney) within 14 days prior to randomization remain within acceptable ranges Willingness of the patient and the sexual partner to use a highly effective contraceptive method during the course of the study
* Able to sufficiently understand the clinical study and give written informed consent

Exclusion Criteria:

* History of major hemorrhage
* High risk of hemorrhage
* History of other malignancies
* Active ulcer
* Patients using anti-coagulants and fibrinolytic drugs
* Active Hepatitis B, or known HBs antigen positive
* Prior treatment history with thrombomodulin alfa
* Administration of another investigational medicinal product within 30 days prior to randomization
* Patient is pregnant (positive urine human chorionic gonadotropin) or breastfeeding or intends to get pregnant during the Treatment period
* Patients otherwise deemed as inappropriate to participate in the study by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Number and Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) | From start of first IMP dose (Cycle 1, Day 1) through End of Treatment (EOT) visit; planned for 6 weeks
  Number and percentage of participants experiencing one or more adverse events which occurred or worsened in severity after the start of the first dose of investigational medicinal product (IMP)
Number and Percentage of Participants with Serious TEAEs | From start of first IMP dose (Cycle 1, Day 1) through EOT visit; planned for 6 weeks
  Number and percentage of participants experiencing one or more serious adverse events which occurred or worsened in severity after the start of the first dose of IMP
Number and Percentage of Participants with TEAEs Leading to Death | From start of first IMP dose (Cycle 1, Day 1) through EOT visit; planned for 6 weeks
  Number and percentage of participants with TEAEs that resulted in death
Number and Percentage of Participants with TEAEs Leading to IMP Discontinuation | From start of first IMP dose (Cycle 1, Day 1) through planned third IMP dose; planned for 4 weeks
  Number and percentage of participants with TEAEs that lead to discontinuation of IMP
Number and Percentage of Participants with Bleeding Events | From start of first IMP dose (Cycle 1, Day 1) through EOT visit; planned for 6 weeks
  Number and percentage of participants experiencing bleeding events
Number and Percentage of Participants with Serious Bleeding Events | From start of first IMP dose (Cycle 1, Day 1) through EOT visit; planned for 6 weeks
  Number and percentage of participants with bleeding events that represent serious adverse events
Number and Percentage of Participants with Dose Limiting Toxicity (DLT) | From start of first IMP dose (Cycle 1, Day 1) until the start of the third IMP dose; planned for 4 weeks
  Number and percentage of participants experiencing DLT
Number and Percentage of Participants with Abnormal Complete Blood Count (CBC) Results | 6 weeks
  Descriptive statistics will summarize the following by cohort: red blood cell count, hemoglobin, hematocrit, white blood cell count, white blood cell differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), and platelet count
Number and Percentage of Participants with Abnormal Serum Chemistry Results | 6 weeks
  Descriptive statistics will summarize the following by cohort: aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase, lactate dehydrogenase, total bilirubin, total protein, albumin, blood urea nitrogen, creatinine, glucose, and electrolytes (sodium, potassium, chloride)
Number and Percentage of Participants with Abnormal Coagulation Panel Results | 6 weeks
  Descriptive statistics will summarize the following by cohort: international normalized ratio (INR), activated partial thromboplastin time (APTT)
Number and Percentage of Participants with Abnormal Qualitative Urinalysis Results | 6 weeks
  Qualitative summary of the following by cohort: protein, glucose, and occult blood
Number and Percentage of Participants with Abnormal Vital Signs | 6 weeks
  Descriptive statistics will summarize the following by cohort: body temperature, pulse, and blood pressure
Number and Percentage of Participants with Anti-ART-123 Antibodies | 6 weeks
  Number and Percentage of Participants with detectable anti-ART-123 antibodies; samples testing positive for anti-ART-123 antibodies will be tested for the presence of neutralizing antibodies

SECONDARY OUTCOMES:
Plasma Concentrations of Thrombomodulin | Cycle 1, Day 1 (each cycle is 14 days)
  Plasma concentrations of thrombomodulin associated with Cycle 1 dosing (each cycle is 14 days)
Plasma Concentrations of 5-fluorouracil (5-FU) | Cycle 1, Day 1 (each cycle is 14 days)
  Plasma concentrations of 5-FU associated with Cycle 1 dosing (each cycle is 14 days)
Plasma Concentrations of Oxaliplatin | Cycle 1, Day 1 and Cycle 3, Day 1 (each cycle is 14 days)
  Plasma concentrations of oxaliplatin associated with Cycle 1 and Cycle 3 dosing (each cycle is 14 days)
Serum Concentrations of Bevacizumab | Cycle 1, Day 1 and Cycle 3, Day 1 (each cycle is 14 days)
  Serum concentrations of bevacizumab associated with Cycle 1 and Cycle 3 dosing (each cycle is 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Libbie McKenzie, MD FASN, Study Director — Veloxis Pharmaceuticals
Locations (32):
- United States (18):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - UCLA Dept. of Medicine - Hematology/Oncology, Los Angeles, California
  - Eastern Connecticut Hematology & Oncology Associates, Norwich, Connecticut
  - Mid-Florida Hematology & Oncology Centers, Orange City, Florida
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - American Oncology Partners, P.A., Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Site #115, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Nashville Oncology Associates, PC, Nashville, Tennessee
  - Site #120, Dallas, Texas
  - Site #114, Houston, Texas
  - MultiCare Regional Cancer Center, Tacoma, Washington
- Japan (14):
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kurashiki Central Hospital, Kurashiki-shi, Okyama
  - NHO Kyushu Cancer Center, Fukuoka
  - Gifu University Hospital, Gifu
  - Kagawa University Hospital, Kita-gun
  - Kitakyushubyoin Kitakyusyu General Hospital, Kitakyushu-shi
  - Kumpukai Sano Hospital, Kobe
  - NHO Shikoku Cancer Center, Matsuyama
  - Kochi Medical School Hospital, Nankoku-shi
  - NHO Osaka National Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Tonan Hospital, Sapporo
  - Shizuoka Cancer Center, Sunto-gun
  - University of Tsukuba Hospital, Tsukuba

IPD SHARING:
Plan to Share IPD: No